CLINICAL TRIAL: NCT04871035
Title: Immunoadsorption Versus Plasma Exchange for Treatment of Guillain-Barré Syndrome (GBS)
Acronym: IPET-GBS
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Collaborators: DiaMed GmbH (Industry)
Responsible Party: Principal Investigator, Albert Christian Ludolph, Prof., Prof. Dr., University of Ulm
Other Study IDs: IPET-GBS 1.2
Record Dates: First submitted 2021-04-28; First posted 2021-05-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: GBS
MeSH Terms: interventions — Plasmapheresis; Plasma Exchange

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunoadsorption
  Interventions: Device: Immunoadsorption
- Plasma Exchange
  Interventions: Device: Plasma Exchange

INTERVENTIONS:
Device: Immunoadsorption — 1 cycle, consisting of 5 sessions on 5 consecutive days with processing of the 0.7-fold individual plasma volume (maximum 2.5 l) each days with tryptophan adsorbers.
  Groups: Immunoadsorption
Device: Plasma Exchange — 1 cycle, consisting of 5 sessions on 5 consecutive days with exchange of 0.7-fold plasma volume (maximum 2.5 l) each day with albumin solution as volume replacement solution.
  Groups: Plasma Exchange

SUMMARY:
This is an observations study evaluating safety and efficacy of immunoadsorption compared to plasma exchange in Guillain-Barré Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Guillain-Barré Syndrome according to the diagnostic criteria proposed by Doorn et al. (Clinical features, pathogenesis, and treatment of Guillain-Barré syndrome, Lancet neurology 2008)
* age 18 years or above

Exclusion Criteria:

* Clinical or laboratory (C-reactive protein 20 mg/l or above, or evidence of nitrite-positive urinary tract infection) evidence of manifest systemic infection
* Intake of angiotensin converting enzyme inhibitor within1 weeks before first treatment
* Other contraindications against immunoadsorption or plasma exchange

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients diagnosed with Guillain-Barré syndrome (GBS) who are treated with either plasma exchange or immunoadsorption in the Department of Neurology, University of Ulm.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2025-05-04 (Estimated); Study Completion 2025-05-04 (Estimated)

PRIMARY OUTCOMES:
Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Score | 2 weeks
  Combined score consisting of Inflammatory Neuropathy Cause and Treatment (INCAT) disability score, Oxford muscle strength score, and vibration score, equally weighted
Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | 2 weeks
  Standard clinical score for inflammatory neuropathies.
Oxford Muscle Strength Score (Medical Research Council, MRC) | 2 weeks
  Standard clinical score for evaluating muscle strength / paresis. Muscle strength will be measured on a scale between 0 (no movement) and 5 (full strength) on 8 pre-defined muscles (one proximal and one distal muscle at each extremity).
Vibration Score | 2 weeks
  Standard clinical score for evaluation of vibration sensitivity on a scale between 0 and 8, using a 256 tuning fork at 4 predefined spots (processus styloideus radii and malleolus lateralis on both sides).

SECONDARY OUTCOMES:
Chronic Inflammatory Demyelinating Polyneuropathy (CIDP) Score | 1, 3, and 5 weeks
  Combined score consisting of Inflammatory Neuropathy Cause and Treatment (INCAT) disability score, Oxford muscle strength score, and vibration score, equally weighted
Inflammatory Neuropathy Cause and Treatment (INCAT) disability score | 1, 3, and 5 weeks
  Standard clinical score for inflammatory neuropathies.
Oxford Muscle Strength Score (Medical Research Council, MRC) | 1, 3, and 5 weeks
  Standard clinical score for evaluating muscle strength / paresis. Muscle strength will be measured on a scale between 0 (no movement) and 5 (full strength) on 8 pre-defined muscles (one proximal and one distal muscle at each extremity).
Vibration Score | 1, 3, and 5 weeks
  Standard clinical score for evaluation of vibration sensitivity on a scale between 0 and 8, using a 256 tuning fork at 4 predefined spots (processus styloideus radii and malleolus lateralis on both sides).
Hughes Score | 1, 2, 3, and 5 weeks
  Standard clinical score to quantify disability in Guillain-Barré syndrome
Pain | 1, 2, 3, and 5 weeks
  Pain quantified on a visual analog scale between 0 (no pain) and 10 (maximum pain).
N20 | 2 and 5 weeks
  N20 latency of nervus medianus (both sides) as measured by somatosensory evoked potentials (SEPs)
P40 | 2 and 5 weeks
  P40 latency of nervus tibialis (both sides) as measured by somatosensory evoked potentials
Nerve Conduction Velocity | 2 and 5 weeks
  Nerve conduction velocity of clinically affected nerves as measured by electroneurography (ENG)
Euro Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) | 1, 2, 3, and 5 weeks
  Quality of Life Scale
Immunoglobulin A in serum | 1, 2, 3, and 5 weeks
  Immunoglobulin A serum concentration
Immunoglobulin A in cerebrospinal fluid (CSF) | 2 weeks
  Immunoglobulin A concentration in cerebrospinal fluid
Immunoglobulin G in serum | 1, 2, 3, and 5 weeks
  Immunoglobulin G serum concentration
Immunoglobulin G in cerebrospinal fluid (CSF) | 2 weeks
  Immunoglobulin G concentration in cerebrospinal fluid
Immunoglobulin M in serum | 1, 2, 3, and 5 weeks
  Immunoglobulin M serum concentration
Immunoglobulin M in cerebrospinal fluid (CSF) | 2 weeks
  Immunoglobulin M concentration in cerebrospinal fluid
Interleukin-1 | 1, 2, 3, and 5 weeks
  Interleukin-1 serum concentration
Interleukin-6 | 1, 2, 3, and 5 weeks
  Interleukin-6 serum concentration
Anti-GM1 antibodies | 1, 2, 3, and 5 weeks
  Anti-GM1 antibody serum levels
Anti-GQ1b | 1, 2, 3, and 5 weeks
  Anti-GQQ1b antibody serum levels
Neurofilament light chain (NfL) serum | 1, 2, 3, and 5 weeks
  Neurofilament light chain (NfL) serum levels
Neurofilament light chain (NfL) in cerebrospinal fluid (CSF) | 2 weeks
  Neurofilament light chain (NfL) levels in cerebrospinal fluid (CSF)
Safety and Tolerability | 1, 2, 3, and 5 weeks
  Kind and frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs)
Therapeutic Response | 1, 2, 3, and 5 weeks
  Share of patients with at least 20% improvement in CIDP score

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Dorst, Prof, Principal Investigator — University of Ulm
Locations (1):
- Department of Neurology, University of Ulm, Ulm, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, and figures), as well as the study protocol will be available. Data will be available beginning 3 months and ending 5 years following article publication. Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal. Proposals should be directed to johannes.dorst@uni-ulm.de; to gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at https://www.uniklinik-ulm.de/neurologie.html.
Supporting Information: Study Protocol
Time Frame: 3 months after publication until 5 years after publication
Access Criteria: Data will be shared with researchers who provide a methodologically sound proposal. Data will be shared for analyses to achieve the aims in the approved proposal.
URL: https://www.uniklinik-ulm.de/neurologie.html